CLINICAL TRIAL: NCT01533116
Title: Effect of BIA 9-1067 at Steady-state on the Pharmacokinetics of a Single-dose of Immediate-release 100/25 mg Levodopa/Carbidopa and 100/25 mg Levodopa/Benserazide in Healthy Subjects
Brief Title: Effect of BIA 9-1067 at Steady-state on the Pharmacokinetics of Levodopa/Carbidopa and Levodopa/Benserazide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BIA-91067-118
Record Dates: First submitted 2012-01-24; First posted 2012-02-15 (Estimated); Results first posted 2015-11-16 (Estimated); Last update posted 2015-11-16 (Estimated); Status verified 2015-10

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; BIA 9-1067
MeSH Terms: conditions — Parkinson Disease | interventions — opicapone; carbidopa, levodopa drug combination; benserazide, levodopa drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 5 mg BIA 9-1067 (Experimental): 5 mg BIA 9-1067 once-daily for 28 days single-dose of levodopa/carbidopa 100/25 mg on Day 21 single-dose of levodopa/benserazide 100/25 mg on Day 28
  Interventions: Drug: BIA 9-1067; Drug: levodopa/carbidopa; Drug: levodopa/benserazide
- Placebo (Experimental): Placebo once-daily for 28 days single-dose of levodopa/carbidopa 100/25 mg on Day 21 single-dose of levodopa/benserazide 100/25 mg on Day 28.
  Interventions: Drug: Placebo; Drug: levodopa/carbidopa; Drug: levodopa/benserazide
- 15 mg BIA 9-1067 (Experimental): 15 mg BIA 9-1067 once-daily for 28 days single-dose of levodopa/carbidopa 100/25 mg on Day 21 single-dose of levodopa/benserazide 100/25 mg on Day 28
  Interventions: Drug: BIA 9-1067; Drug: levodopa/carbidopa; Drug: levodopa/benserazide
- 30 mg BIA 9-1067 (Experimental): 30 mg BIA 9-1067 once-daily for 28 days single-dose of levodopa/carbidopa 100/25 mg on Day 21 single-dose of levodopa/benserazide 100/25 mg on Day 28
  Interventions: Drug: BIA 9-1067; Drug: levodopa/carbidopa; Drug: levodopa/benserazide

INTERVENTIONS:
Drug: BIA 9-1067
  Other Names: OPC, Opicapone
  Arms: 15 mg BIA 9-1067; 30 mg BIA 9-1067; 5 mg BIA 9-1067
Drug: Placebo
  Other Names: PLC, Placebo
  Arms: Placebo
Drug: levodopa/carbidopa
  Other Names: Sinemet® 100/25
Drug: levodopa/benserazide
  Other Names: Prolopa® 100/25

SUMMARY:
To investigate the effect of BIA 9-1067 in steady-state conditions on the levodopa pharmacokinetics

DETAILED DESCRIPTION:
Single centre, randomized, double-blind, gender-balanced, placebo-controlled study in 4 groups of healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Availability for the entire study period and willingness to adhere to the protocol requirements as evidenced by the informed consent form (ICF) duly read, signed and dated by the volunteer prior to participation in the study.
* Male or female volunteers.
* Volunteers of at least 25 years of age but not older than 45 years.
* Volunteers with body mass index (BMI) greater than or equal to 19 and below 30 kg/m2.
* Volunteers who were healthy as determined by pre-study (at screening) medical history, physical examination, vital signs, complete neurological examination and 12-lead ECG.
* Volunteers who had clinical laboratory test results judged clinically acceptable (within the laboratory's stated normal range; if not within this range, they must had been without any clinical significance) at screening and admission to first treatment period.
* Volunteers who had negative tests for hepatitis B surface antigen (HBsAg), anti-hepatitis C antibodies (HCV Ab), and Human immunodeficiency viruses -1 and -2 antibodies (HIV-1 and HIV-2 Ab) at screening.
* Volunteers who had negative screen of ethyl alcohol and drugs of abuse at screening and admission to the treatment period.
* Volunteers who were non- or ex-smokers. For the purpose of this study, an ex-smoker is defined as someone who completely stopped smoking for at least 3 months before day 1 of this study.
* Due to unknown risks and potential harm to the unborn fetus, sexually active men or women must have agreed to use a medically acceptable form of contraception throughout the study.
* If female of childbearing potential, she had a negative HCG beta serum pregnancy test at screening and admission to each treatment period.
* The informed consent form must have been signed by all volunteers, prior to their participation in the study.

Exclusion Criteria:

* Volunteers who did not conform to the above inclusion criteria, or in case of
* Volunteers who had a clinically relevant surgical history.
* Volunteers who had a clinically relevant family history.
* Volunteers who had a history of relevant atopy.
* Volunteers who had a significant infection or known inflammatory process at screening or admission to the treatment period.
* Volunteers who had acute gastrointestinal symptoms at the time of screening or admission to the treatment period (e.g., nausea, vomiting, diarrhoea, heartburn).
* Volunteers who were vegetarians, vegans or have medical dietary restrictions.
* Volunteers who could not communicate reliably with the investigator.
* Volunteers who were unlikely to co-operate with the requirements of the study.
* History of hypersensitivity to BIA 9-1067, tolcapone, entacapone, levodopa, benserazide or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs.
* Presence of significant gastrointestinal, liver or kidney disease, or any other conditions known to interfere with the absorption, distribution, metabolism or excretion of drugs or known to potentiate or predispose to undesired effects.
* History of significant gastrointestinal, liver or kidney disease that may affect drug bioavailability.
* Presence or history of significant cardiovascular, pulmonary, hematologic, neurologic, psychiatric, lymphatic, musculoskeletal, genitourinary, endocrine, immunologic, dermatologic or connective tissue disease.
* Suicidal tendency, history of or disposition to seizures, state of confusion, clinically relevant psychiatric diseases.
* Presence of significant heart disease or disorder according to ECG.
* Presence of suspicious undiagnosed skin lesions or a history of melanoma.
* Previous history of Neuroleptic Malignant Syndrome (NMS) and/or nontraumatic rhabdomyolysis.
* History of significant glaucoma.
* Used of prescription medications including monoamine oxidase (MAO) inhibitors within 28 days before day 1 of the study.
* Used of over-the-counter (OTC) products within 7 days before day 1 of the study.
* Maintenance therapy with any drug, or significant history of drug dependency (drug abuse) or alcohol abuse (> 3 units of alcohol per day, intake of excessive alcohol, acute or chronic).
* Any clinically significant illness in the previous 28 days before day 1 of this study.
* Volunteers who took an Investigational Product (in another clinical trial) or donated 50 mL or more of blood in the previous 28 days before day 1 of this study.
* Poor motivation, intellectual problems likely to limit the validity of consent to participate in the study or limit the ability to comply with the protocol requirements or inability to cooperate adequately, inability to understand and to observe the instructions of the physician.
* Donation of 500 mL or more of blood (Canadian Blood Services, Hema-Quebec, clinical studies, etc.) in the previous 56 days before day 1 of this study.
* Positive urine screening of ethyl alcohol or drugs of abuse at admission to the treatment period.
* Any history of tuberculosis and/or prophylaxis for tuberculosis.
* Positive results to HIV, HBsAg or anti-HCV tests.
* Participation in any previous clinical study with BIA 9-1067.
* Females who were pregnant according to a positive serum pregnancy test or were lactating.
* Females of childbearing potential who refused to use an acceptable contraceptive regimen throughout the study.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2009-03; Primary Completion 2009-08 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sicard, MD, Principal Investigator — Algorithme Pharma Inc
Locations (1):
- Algorithme Pharma Inc., Mount Royal, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo once-daily for 28 days single-dose of levodopa/carbidopa 100/25 mg on Day 21 single-dose of levodopa/benserazide 100/25 mg on Day 28.
  Placebo
  levodopa/carbidopa
  levodopa/benserazide
- 5 mg BIA 9-1067: 5 mg BIA 9-1067 once-daily for 28 days single-dose of levodopa/carbidopa 100/25 mg on Day 21 single-dose of levodopa/benserazide 100/25 mg on Day 28
  BIA 9-1067
  levodopa/carbidopa
  levodopa/benserazide
- 15 mg BIA 9-1067: 15 mg BIA 9-1067 once-daily for 28 days single-dose of levodopa/carbidopa 100/25 mg on Day 21 single-dose of levodopa/benserazide 100/25 mg on Day 28
  BIA 9-1067
  levodopa/carbidopa
  levodopa/benserazide
- 30 mg BIA 9-1067: 30 mg BIA 9-1067 once-daily for 28 days single-dose of levodopa/carbidopa 100/25 mg on Day 21 single-dose of levodopa/benserazide 100/25 mg on Day 28
  BIA 9-1067
  levodopa/carbidopa
  levodopa/benserazide
Period: Overall Study
Arm/Group | Placebo | 5 mg BIA 9-1067 | 15 mg BIA 9-1067 | 30 mg BIA 9-1067
Started | 14 | 13 | 13 | 12
Completed | 12 | 12 | 12 | 12
Not Completed | 2 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 5 mg BIA 9-1067 | 15 mg BIA 9-1067 | 30 mg BIA 9-1067 | Total
Number analyzed (Participants) | 14 | 13 | 13 | 12 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 13 | 13 | 12 | 52
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 6 | 6 | 25
  Male | 7 | 7 | 7 | 6 | 27

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Plasma Concentration
Description: Cmax - maximum plasma concentration Cmax (Levodopa) Sinemet® or Prolopa® - following administration of Sinemet® or Prolopa® Cmax (3-OMD) Sinemet® or Prolopa® - following administration of Sinemet® or Prolopa® Cmax (BIA 9-1067) Sinemet® or Prolopa® - following administration of Sinemet® or Prolopa®
Time Frame: pre-dose and at the following times post-dose: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 h
Population: According to the protocol, the "pharmacokinetic population" should include all subjects who had valid levodopa pharmacokinetic data. In this study, 48 subjects completed the entire study and 49 had valid levodopa data (one subject had valid levodopa data until Day 21)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo | 5 mg BIA 9-1067 | 15 mg BIA 9-1067 | 30 mg BIA 9-1067
Number analyzed (Participants) | 13 | 12 | 12 | 12
ng/mL
  Cmax (Levodopa) Sinemet® 100/25 | 985 (290) | 1245 (524) | 1200 (607) | 944 (256)
  Cmax (Levodopa) Prolopa® 100-25 | 1704 (682) | 2100 (907) | 1727 (957) | 1795 (788)
  Cmax (3-OMD) Sinemet® 100/25 | 456 (130) | 307 (106) | 167 (82.5) | 115 (54.5)
  Cmax (3-OMD) Prolopa® 100/25 | 688 (230) | 360 (96) | 206 (110.8) | 160 (61.9)
  Cmax (BIA 9-1067) Sinemet® 100/25 | NA (NA) — BIA 9-1067 was not administered | 75.0 (39) | 263 (82.3) | 310 (115)
  Cmax (BIA 9-1067) Prolopa® 100/25 | NA (NA) — BIA 9-1067 was not administered | 95.5 (41.1) | 281 (153.4) | 370 (181.7)

2. Primary Outcome: Tmax - Time to Maximum Plasma Concentration
Description: Tmax - time to maximum plasma concentration Tmax (Levodopa) Sinemet® or Prolopa® - following administration of Sinemet® or Prolopa® Tmax (3-OMD) Sinemet® or Prolopa® - following administration of Sinemet® or Prolopa® Tmax (BIA 9-1067) Sinemet® or Prolopa® - following administration of Sinemet® or Prolopa®
Time Frame: pre-dose and at the following times post-dose: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 h
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Placebo | 5 mg BIA 9-1067 | 15 mg BIA 9-1067 | 30 mg BIA 9-1067
Number analyzed (Participants) | 13 | 12 | 12 | 12
hours
  Tmax (Levodopa) Sinemet® 100/25 | 0.5 [0.5 to 3.0] | 0.75 [0.5 to 3.0] | 0.5 [0.5 to 1.5] | 1.0 [0.5 to 2.0]
  Tmax (Levodopa) Prolopa® 100-25 | 1.0 [0.5 to 2.0] | 1.0 [0.5 to 1.5] | 1.0 [0.5 to 2.0] | 1.0 [0.5 to 2.0]
  Tmax (3-OMD) Sinemet® 100/25 | 4.0 [4.0 to 6.0] | 8.0 [6.0 to 8.0] | 6.0 [3.0 to 8.0] | 8.0 [4.0 to 8.0]
  Tmax (3-OMD) Prolopa® 100/25 | 4.0 [3.0 to 6.0] | 8.0 [4.0 to 8.0] | 6.0 [2.0 to 8.0] | 4.0 [3.0 to 8.0]
  Tmax (BIA 9-1067) Sinemet® 100/25 | NA [NA to NA] — BIA 9-1067 was not administered | 1.5 [0.5 to 6.0] | 3.0 [1.5 to 6.0] | 4.0 [1.5 to 6.0]
  Tmax (BIA 9-1067) Prolopa® 100/25 | NA [NA to NA] — BIA 9-1067 was not administered | 3.0 [1.0 to 4.0] | 2.5 [0.5 to 6.0] | 3.0 [1.0 to 6.0]

3. Primary Outcome: AUC0-t - Area Under the Plasma Concentration-time Curve to Last Measurable Time Point
Description: AUC0-t - area under the plasma concentration-time curve from time 0 to last observed concentration 3-OMD - 3-O-methyl-dopa - metabolite of L-DOPA (levodopa) AUC0-t (Levodopa) Sinemet® or Prolopa® - following administration of Sinemet® or Prolopa® AUC0-t (3-OMD) Sinemet® or Prolopa® - following administration of Sinemet® or Prolopa® AUC0-t (BIA 9-1067) Sinemet® or Prolopa® - following administration of Sinemet® or Prolopa®
Time Frame: pre-dose and at the following times post-dose: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 h
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Placebo | 5 mg BIA 9-1067 | 15 mg BIA 9-1067 | 30 mg BIA 9-1067
Number analyzed (Participants) | 13 | 12 | 12 | 12
ng.h/mL
  AUC0-t (Levodopa) Sinemet® 100/25 | 1837 (593) | 3386 (1449) | 2952 (1003) | 2753 (889)
  AUC0-t (Levodopa) Prolopa® 100-25 | 2438 (712) | 4115 (1547) | 3442 (1225) | 4056 (1051)
  AUC0-t (3-OMD) Sinemet® 100/25 | 7631 (1786) | 5147 (1534) | 2836 (1495) | 1751 (988)
  AUC0-t (3-OMD) Prolopa® 100/25 | 11371 (3707) | 6205 (1458) | 3473 (1962) | 2623 (1065)
  AUC0-t (BIA 9-1067) Sinemet® 100/25 | NA (NA) — BIA 9-1067 was not administered | 223 (58.2) | 872 (412) | 1101 (525)
  AUC0-t (BIA 9-1067) Prolopa® 100/25 | NA (NA) — BIA 9-1067 was not administered | 232 (82.4) | 836 (497) | 1185 (562)

4. Primary Outcome: tEmax - Time of Occurrence of Maximum Observed Effect on S-COMT Activity
Description: tEmax - time of occurrence of maximum observed effect on S-COMT activity COMT - Catechol-O-Methyltransferase
Time Frame: pre-dose and at the following times post-dose: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 h
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Placebo | 5 mg BIA 9-1067 | 15 mg BIA 9-1067 | 30 mg BIA 9-1067
Number analyzed (Participants) | 13 | 12 | 12 | 12
hours | 8.12 (8.15) | 2.71 (2.16) | 4.67 (1.92) | 3.50 (2.41)

5. Primary Outcome: AUEC0-24 - Area Under the Effect-time Curve (AUEC) to 24 h Post-dose
Description: AUEC0-24 - Area under the effect-time curve (AUEC) to 24 h post-dose.
Time Frame: pre-dose and at the following times post-dose: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 h
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pmol/mg Hb/h.h
Arm/Group | Placebo | 5 mg BIA 9-1067 | 15 mg BIA 9-1067 | 30 mg BIA 9-1067
Number analyzed (Participants) | 13 | 12 | 12 | 12
pmol/mg Hb/h.h | 906 (276) | 454 (97.3) | 319 (134) | 226 (177)

ADVERSE EVENTS:
Arm/Group | Placebo | 5 mg BIA 9-1067 | 15 mg BIA 9-1067 | 30 mg BIA 9-1067
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13 | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 11/14 | 9/13 | 11/13 | 9/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=14) | 5 mg BIA 9-1067 (N=13) | 15 mg BIA 9-1067 (N=13) | 30 mg BIA 9-1067 (N=12)
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Dark circles under eyes (Eye disorders) | 0 | 0 | 1 | 0
Eye pain (Eye disorders) | 0 | 0 | 1 | 0
Eye pruritus (Eye disorders) | 1 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 1 | 1 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 2 | 1
Eructation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 1 | 1
Chest discomfort (General disorders) | 0 | 0 | 0 | 1
Chills (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 2 | 1
Feeling hot (General disorders) | 0 | 0 | 0 | 1
Vessel puncture site reaction (General disorders) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Sunburn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Blood potassium increased (Investigations) | 0 | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 2
Dizziness (Nervous system disorders) | 2 | 3 | 1 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 1 | 1 | 3
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Sensory disturbance (Nervous system disorders) | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 5 | 3 | 5 | 6
Euphoric mood (Psychiatric disorders) | 1 | 0 | 0 | 0
Polyuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urine odour abnormal (Renal and urinary disorders) | 1 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Hot flush (Vascular disorders) | 1 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other